CLINICAL TRIAL: NCT06391931
Title: A Multicenter, Open, Controlled, Phase III Clinical Study to Evaluate the Efficacy and Safety of Cipepofol Injection for General Anesthesia in Pediatric Patients Undergoing Elective Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-310
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cipepofol group (Experimental)
  Interventions: Drug: Cipepofol
- Propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Cipepofol — 0.6±0.2 mg/kg induce + 0.8 mg/kg/h maintain
  Arms: Cipepofol group
Drug: Propofol — 3.0 mg/kg induce + 5.0 mg/kg/h maintain
  Arms: Propofol group

SUMMARY:
A multicenter, open, controlled, Phase III clinical study to evaluate the efficacy and safety of Cipepofol injection for general anesthesia in pediatric patients undergoing elective surgery

ELIGIBILITY:
Inclusion Criteria:

* Age ≥2 years old and < 18 years old, gender is not limited;
* Selective surgery requiring tracheal intubation, mechanical ventilation and general anesthesia, with an estimated anesthetic time of 30 to 120 minutes;
* Intravenous anesthesia is suitable for both induction and maintenance of general anesthesia;
* ASA grade I-II;
* Before any activities related to the trial, the child's guardian or his/her guardian should sign the informed consent.

Exclusion Criteria:

* The type of operation is emergency rescue operation or emergency rescue is required during the operation or blood transfusion may be required according to the researchers;
* Patients with contraindications to general anesthesia or who have a history of anesthesia accidents;
* Known or suspected allergy to excipients in propofol injection, Cipepofol injection excipients (soybean oil, glycerol, triglyceride, yolk lecithin, sodium oleate and sodium hydroxide), benzodiazepines, opioids, rocuronium bromide, atropine, etc., and their active ingredients; Contraindications of propofol injection;
* Prior to screening/baseline, the following medical history or evidence of increased risk of sedation/anesthesia was collected and was determined by the investigator to be inappropriate: Cardiovascular system diseases: severe congenital heart disease (such as tetralogy of Fallot, etc.), severe arrhythmias (such as tachycardia/bradycardia requiring medical treatment, degree III atrioventricular block), severe heart failure, etc.; Respiratory diseases: respiratory insufficiency, history of bronchospasm/asthma requiring treatment within 1 month prior to screening, acute upper respiratory infection with obvious fever, wheezing, or phlegm-producing cough within 1 week prior to baseline; Craniocerebral diseases: history of craniocerebral injury, convulsion, epilepsy, intracranial hypertension, cerebral aneurysm, cerebrovascular accident; Or a known history of mental disorders, such as seizures, schizophrenia, mania, long-term use of psychiatric drugs, cognitive dysfunction; Gastrointestinal diseases: gastrointestinal retention, active bleeding, may lead to reflux aspiration and other conditions; a history of uncontrolled, clinically significant disease of the liver, kidney, hematological, nervous, or metabolic system; Patients with severe infection, trauma or major surgical operation within 4 weeks prior to screening; A history or family history of malignant hyperthermia.
* There are any of the following respiratory management risks within 1 week before screening: Asthma attacks, wheezing; Patients with failed tracheal intubation experience; The investigators assessed the risk of difficulty with mask ventilation or intubation.
* Participants who have participated in any drug clinical trial within 1 month before screening;
* Laboratory examination indicators in the screening period/baseline period meet the following standards and are confirmed by review: alanine aminotransferase and/or ASpartate aminotransferase ≥ 5.0× Upper limit of normal (ULN); Total bilirubin ≥3.0×ULN; serum creatinine ≥2.5×ULN.
* Women who are fertile (i.e. post-menarche) and do not wish to use contraception throughout the trial period;
* Paediatric population requiring special care or supervision by courts/social welfare institutions;
* Subjects who have any other factors deemed unsuitable by the investigator for participation in this study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Success rate of anesthesia | 24 hours after the end of surgery
  Success rate of anesthesia induction and anesthesia maintenance

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No